CLINICAL TRIAL: NCT03797846
Title: Comparison of Effectiveness and Safety of Eye Fixation Types During Combined Glaucoma Procedures
Brief Title: Comparison of Fixation Suture Type in Glaucoma Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Joanna Konopińska, MD, PhD, Medical University of Bialystok
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1771
Record Dates: First submitted 2019-01-03; First posted 2019-01-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Glaucoma Eye; Glaucoma
Keywords: ptosis; combined procedures; glaucoma; post-surgery complication
MeSH Terms: conditions — Glaucoma; Blepharoptosis

STUDY DESIGN:
Intervention Model Description: A prospective randomized trial with a 6 month follow-up period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corneal Suture (Active Comparator): intraoperative fixation with the suture in clear cornea qualified to the combined glaucoma surgery
  Interventions: Procedure: combined glaucoma surgery
- Muscle Suture (Active Comparator): intraoperative fixation with the bridle suture for superior rectus muscle qualified to the combined glaucoma surgery
  Interventions: Procedure: combined glaucoma surgery

INTERVENTIONS:
Procedure: combined glaucoma surgery — combined procedure with trabeculectomy and cataract removal

SUMMARY:
The aim of the study is to compare the effectiveness and safety of two types of intraoperative eye fixation: for the superior rectus muscle and traction suture in the peripheral cornea.

This is a prospective randomized trial with a 6 month follow-up period, which covers patients with open angle glaucoma qualified for combined glaucoma procedure (phacotrabeculectomy). In I group, the intraoperatively fixation in the peripheral part of the cornea is used, in II group the bridle suture for the superior rectus muscle is performed.

DETAILED DESCRIPTION:
The way of the intraoperatively fixation may have some impact for postoperative results of the level of intraocular pressure (IOP), visual acuity (BCVA) and the incidence of upper eyelid ptosis was determined as a post-operative MRD (margin reflex distance) ≥2mm.

ELIGIBILITY:
Inclusion Criteria:

* co-existing glaucoma and cataract (NC1, NC2) classified by means of the LOCS III scale (Lens Opacities Classification System III)
* primary open-angle glaucoma and secondary pseudoexfoliative glaucoma, in which a satisfactory IOP level was not achieved despite maximum tolerable hypotensive treatment, both topical and systemic
* documented progression of loss of field of vision
* significant daily IOP fluctuations
* no cooperation from patient with regard to application of anti-glaucoma treatment, allergy to topical medications

Exclusion Criteria:

* no consent to participation in the study
* prior surgical and laser procedures in the area of the eye
* narrow- or closed-angle glaucoma
* post-inflammatory or post-traumatic secondary glaucoma
* chronic illness of the cornea or optic nerve
* advanced macular degeneration
* active inflammatory process
* pregnancy
* systemic steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
IOP | baseline and twelve months after surgery
  the change in the level of intraocular pressure

SECONDARY OUTCOMES:
BCVA | baseline and twelve months after surgery
  the change in the best corrected visual acuity
MRD | baseline and twelve months after surgery
  the incidence of upper eyelid ptosis determined as a post-operative MRD (margin reflex distance) ≥2mm

CONTACTS AND LOCATIONS:
Overall Officials: Zofia Mariak, Prof, Study Chair — Medical University of Bialystok
Locations (1):
- Medical University, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of each participant will be available on email request for all primary and secondary outcome measures
Supporting Information: Study Protocol
Time Frame: Data will be available on email request for six months after completing recruitment
Access Criteria: e-mail request, after Data Access Agreement is sign

REFERENCES:
- [Background] Li B, Zhang M, Liu W, Wang J. Comparison of Superior Rectus and Peripheral Lamellar Corneal Traction Suture during Trabeculectomy. Curr Eye Res. 2016;41(2):215-21. doi: 10.3109/02713683.2015.1009635. Epub 2015 Sep 15. PMID 25803293